CLINICAL TRIAL: NCT04518215
Title: Ultrasound-Guided Erector Spinae Plane Block for Paediatric Upper Abdominal Surgery: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block for Paediatric Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USESPBPUAS
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Paediatric; Surgery; Analgesia; Anesthesia
Keywords: Erector spinae plain block; Ultrasound-guided; Paediatric; Upper abdominal surgery; Analgesia; Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Experimental): Erector Spinae Plain Block
  Interventions: Procedure: Erector Spinae Plain Block; Procedure: Intra-Venous Analgesia
- IV Analgesia group (Active Comparator): Intra-Venous Analgesia
  Interventions: Procedure: Intra-Venous Analgesia

INTERVENTIONS:
Procedure: Erector Spinae Plain Block — Patients will receive erector spinae plane block (ESP) at the level of T 9-10. Following skin sterilization, high-frequency linear ultrasound probe will be placed 1-2 cm lateral to the midline at the T 9 level. After identification of the erector spinae muscle (ESM) and the transverse process; a 22 G needle will be inserted, in a cranio-caudal direction, deep into the ESM in an in-plane technique. Correct needle placement will be verified with the administration of 0.5-1 ml Normal Saline to view the hydrodissection between the transverse process and the ESM. 0.25% Bupivacaine in a calculated volume of 0.5 ml/kg (with a maximum dose of 20 ml) will be injected deep to the erector spinae muscle for unilateral ESPB.
  Arms: ESPB group
Procedure: Intra-Venous Analgesia — Post-operative rescue analgesic plan will consist of 15 mg/kg Paracetamol IV if the FLACC [Face, Leg, Activity, Cry, Consolability] score is 2-4 and 1 mg/kg Tramadol IV if FLACC score > 4.

SUMMARY:
Upper abdominal surgeries are associated with severe postoperative pain. Thus, maintaining effective postoperative analgesia in the paediatric age group is very crucial in terms of future pain perception and chronic pain development. Erector Spinae Plane Block (ESPB) is an interfascial plane block characterized by its ease of application and low complication rates with the introduction of ultrasonography. The aim of this study is to investigate the analgesic effects of ESPB in this particular age-group.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II.
* Elective open upper abdominal surgeries, e.g., open cholecystectomy, splenectomy, pyeloplasty, renal cysts excision, partial or total nephrectomy.

Exclusion Criteria:

* Patient's next of kin refusal.
* Allergy to local anaesthetics.
* Infection at the site of injection.
* Coagulopathy.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Tramadol consumption. | 24 hours
  Total dose of Tramadol (measured in mg) given intra-venously to the patient post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Atef K Salama, MD, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Nazmy S Michael, MD, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided